CLINICAL TRIAL: NCT00372827
Title: Efficacy and Safety of Timolol Maleate 0.5% Compared to Brinzolamide 1% When Added to Travoprost 0.004% in Primary Open-angle Glaucoma or Ocular Hypertension
Brief Title: Study of Brinzolamide and Timolol When Added to Travoprost in Primary Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-03-06
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2008-05

CONDITIONS: Primary Open-angle Glaucoma; Ocular Hypertension; Pigment Dispersion Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide

INTERVENTIONS:
Drug: Brinzolamide 1% added to Travoprost 0.004%

SUMMARY:
The purpose of the study is to compare the efficacy and safety of Timolol 0.5% solution to Brinzolamide 1% each given twice daily when added to Travoprost 0.004% given each evening.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated with any prostaglandin analogue monotherapy (excluding unoprostone) and who have an intraocular pressure between 19 and 32 mmHg at 08:00 hours.

Exclusion Criteria:

* Under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245
Dates: Start 2004-02; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Mean diurnal intraocular pressure at month 3

SECONDARY OUTCOMES:
Individual intraocular pressures measured at 08:00, 12:00 and 16:00 at month 3.
Reduction from baseline in mean diurnal intraocular pressure and individual timepoints.
Visual acuity, Slit lamp biomicroscopy and adverse events during 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Grau, Study Director — Study Manager
Locations (1):
- Mainz Site, Mainz, Germany

REFERENCES:
- [Result] Hollo G, Chiselita D, Petkova N, Cvenkel B, Liehneova I, Izgi B, Berta A, Szaflik J, Turacli E, Stewart WC. The efficacy and safety of timolol maleate versus brinzolamide each given twice daily added to travoprost in patients with ocular hypertension or primary open-angle glaucoma. Eur J Ophthalmol. 2006 Nov-Dec;16(6):816-23. doi: 10.1177/112067210601600606. PMID 17191187